CLINICAL TRIAL: NCT02632851
Title: Non-interventional Multicentric Study on Treatment of Respiratory Tract Infection and/or Acute Bronchitis With Ectoin Inhalation Solution
Brief Title: Treatment of Respiratory Tract Infection and/or Acute Bronchitis With Ectoin Inhalation Solution
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: EIL/aBr/2015
Record Dates: First submitted 2015-12-02; First posted 2015-12-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Bronchitis; Cough; Sputum, Cellular Atypia; Dyspnoea
Keywords: inhalation; isotonic saline; NaCl solution 0.9 %; Ectoin; bronchitis; respiratory tract infection
MeSH Terms: conditions — Bronchitis; Cough; Dyspnea; Respiratory Aspiration; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ectoin inhalation solution: treatment according to instructions for use
- Pari NaCl inhalation solution (0.9%): treatment according to instructions for use

SUMMARY:
This observational, non-interventional multicentric study compares the inhalation therapy on patients suffering on respiratory tract infections and/or acute bronchitis between Ectoin inhalation solution and Pari NaCl (0.9%) inhalation solution

DETAILED DESCRIPTION:
The assessment focuses on the bronchitis Severity Score (BSS) for standardized use in clinical studies with the outcome criteria of cough, sputum production, rales/rhonchi, chest pain during coughing and dysnoea

ELIGIBILITY:
Inclusion Criteria:

* according to instruction for use

Exclusion Criteria:

* according to instruction for use

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care or ENT units study the therapeutic process in this obvservational trial in total of 120 patients suffering on respiratory tract infection and/or acute bronchitis
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Bronchitis Severity Score on physician´s evaluation (5 point IMOS scale) | day 7
  Assessment of bronchits severity score on a 5 point IMOS scale (complete recovery, major improvement, slight to moderate improvement, no change, deterioration) of symptoms:
  Cough, sputum production, rales/rhonchi, chest pain during coughing, dyspnoea

SECONDARY OUTCOMES:
Change in bronchitis symptoms evaluated on patients´ diaries (5 point scale) | day 14
  Assessment of bronchits symptoms on a 5 point scale (absent, mild, moderate, severe, very severe) of symptoms:
  Cough, sputum production, rales/rhonchi, chest pain during coughing, dyspnoea
patients´ evaluation of tolerability (4 point scale) | day7
  assessment of tolerability on a 4 point scale (bad, satisfied, good, very good)
physicians´ evaluation of tolerability (4 point scale) | day 7
  assessment of tolerability on a 4 point scale (bad, satisfied, good, very good)
patients´ evaluation of efficacy (five point IMOS scale) | day 7
  assessment of tolerability on a five point IMOS scale (complete recovery, major improvement, slight to moderate improvement, no change, deterioration)
physicians´ evaluation of efficacy (five point IMOS scale) | day 7
  assessment of tolerability on a five point IMOS scale (complete recovery, major improvement, slight to moderate improvement, no change, deterioration)
Change in number and type of adverse events | day 7
  incidence of adverse events and correlation with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: R Mösges, Prof Dr, Study Chair — University of Cologne
Locations (1):
- Facharzt für HNO, Allergologie, Cologne, Germany

REFERENCES:
- [Background] Matthys H, Kamin W. Positioning of the Bronchitis Severity Score (BSS) for standardised use in clinical studies. Curr Med Res Opin. 2013 Oct;29(10):1383-90. doi: 10.1185/03007995.2013.832183. Epub 2013 Aug 23. PMID 23927521